CLINICAL TRIAL: NCT00392847
Title: Promoting Parental Skills and Enhancing Attachment in Early Childhood
Acronym: CAPEDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: P051045
Record Dates: First submitted 2006-10-17; First posted 2006-10-26 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Behavioral Disorders
Keywords: Child mental disorder; Home visit; Postnatal depression; Social Support; Random selection
MeSH Terms: conditions — Mental Disorders; Neurodevelopmental Disorders; Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): The first group will receive routine follow-up as currently provided by national community health and social services.
  Interventions: Behavioral: Promoting Parental Skills and Enhancing Attachment
- 1 (Experimental): will receive home visits by community workers. These visits will start during pregnancy and will continue up to the child's second birthday.
  Interventions: Behavioral: had home visits by community workers during pregnancy

INTERVENTIONS:
Behavioral: Promoting Parental Skills and Enhancing Attachment — The first group will receive routine follow-up as currently provided by national community health and social services.
  Arms: 2
Behavioral: had home visits by community workers during pregnancy — had home visits by community workers during pregnancy to the child's second birthday.
  Other Names: to the child's second birthday.
  Arms: 1

SUMMARY:
Child psychological/behavioural disorders such as withdrawal may persist when the psychosocial context is unfavourable. Health promotion strategies (Olds' paradigm) have proved their efficacy in vulnerable populations. CAPEDP project sets out to evaluate a program of home visits in France

DETAILED DESCRIPTION:
This program aims at reducing psychosocial disorders and promoting mental health, social support and attachment amongst at-risk young women and their family. 440 primigravida (pregnant women) will be randomised into two groups. The first group will receive routine follow-up as currently provided by national community health and social services. The second group will receive home visits by community workers. These visits will start during pregnancy and will continue up to the child's second birthday.

ELIGIBILITY:
Inclusion Criteria:

* Being less than 26 years old
* Being pregnant for less than 27 weeks
* Being primiparous
* Living in the study area
* Being socially vulnerable: less than 12 years of education AND/OR socially isolated AND/OR eligible for a public health insurance for people with low resources.

Exclusion Criteria:

* Refusal to participate
* Not able to speak French
* Having a medical follow-up which necessitates regular contact with health professional
* Not having health insurance
* Persons for whom follow up at 27 months is impossible (evaluation at baseline)

Max Age: 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 440 (Actual)
Dates: Start 2006-12; Primary Completion 2011-08 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Mothers' scores on a postnatal depression scale (baseline, and when the child is 3, 6 and 12 months old) | baseline, and when the child is 3, 6 and 12 months old
Parental competencies (when the child is 3, 12 and 18 months old) | when the child is 3, 12 and 18 months old
Child mental health (when the child is 18 and 24 months old) | when the child is 18 and 24 months old

SECONDARY OUTCOMES:
Child attachment (when the child is 18 months old) | when the child is 18 months old
Family use of medical and social services (baseline, and when the child is 3, 6, 12 and 24 months old) | baseline, and when the child is 3, 6, 12 and 24 months old
Family social support (baseline, and when the child is 3, 12 and 24 months old) | baseline, and when the child is 3, 12 and 24 months old
Mother's self-esteem as a parent (when the child is 3, 12 and 24 months old) | when the child is 3, 12 and 24 months old
Child psychomotor development (when the child is 6, 12 and 24 months old) | when the child is 6, 12 and 24 months old
Mother's knowledge about child development (baseline, and when the child is 3 and 24 months old) | baseline, and when the child is 3 and 24 months old
Mother's attachment (at baseline) | at baseline
Mother's mental health (baseline, and when the child is 3 and 24 months old) | baseline, and when the child is 3 and 24 months old
Mother's working alliance with home visitor (not for control group) (when the child is 3, 6, 12 and 24 months old) | not for control group,when the child is 3, 6, 12 and 24 months old
Social-demographic data (all follow-up points: baseline, and when the child is 3, 6, 12, 18 and 24 months old) | baseline, and when the child is 3, 6, 12, 18 and 24 months old

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Guedeney, PU-PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Bichat-Claude Bernard Hospital, Paris, France

REFERENCES:
- [Result] Dugravier R. [Understanding consequences of hospitalization within attachment theory]. Arch Pediatr. 2010 Jun;17(6):723-4. doi: 10.1016/S0929-693X(10)70078-6. No abstract available. French. PMID 20654860
- [Result] Guedeney A, Guedeney N, Tereno S, Dugravier R, Greacen T, Welniarz B, Saias T, Tubach F; CAPEDP Study Group. Infant rhythms versus parental time: promoting parent-infant synchrony. J Physiol Paris. 2011 Dec;105(4-6):195-200. doi: 10.1016/j.jphysparis.2011.07.005. Epub 2011 Jul 12. PMID 21782020
- [Result] Saias T, Lerner E, Greacen T, Simon-Vernier E, Emer A, Pintaux E, Guedeney A, Dugravier R, Tereno S, Falissard B, Tubach F; CAPEDP Study Group; Revah-Levy A. Evaluating fidelity in home-visiting programs a qualitative analysis of 1058 home visit case notes from 105 families. PLoS One. 2012;7(5):e36915. doi: 10.1371/journal.pone.0036915. Epub 2012 May 18. PMID 22629341
- [Derived] Greacen T, Welniarz B, Purper-Ouakil D, Wendland J, Dugravier R, Saias T, Tereno S, Tubach F, Haddad A, Guedeney A; CAPEDP STUDY GROUP. BEST PRACTICE IN INDIVIDUAL SUPERVISION OF PSYCHOLOGISTS WORKING IN THE FRENCH CAPEDP PREVENTIVE PERINATAL HOME-VISITING PROGRAM: RESULTS OF A DELPHI CONSENSUS PROCESS. Infant Ment Health J. 2017 Mar;38(2):267-275. doi: 10.1002/imhj.21630. Epub 2017 Feb 25. PMID 28236309
- [Derived] Dugravier R, Tubach F, Saias T, Guedeney N, Pasquet B, Purper-Ouakil D, Tereno S, Welniarz B, Matos J; CAPEDP Study Group; Guedeney A, Greacen T. Impact of a manualized multifocal perinatal home-visiting program using psychologists on postnatal depression: the CAPEDP randomized controlled trial. PLoS One. 2013 Aug 19;8(8):e72216. doi: 10.1371/journal.pone.0072216. eCollection 2013. PMID 23977257
- [Derived] Tubach F, Greacen T, Saias T, Dugravier R, Guedeney N, Ravaud P, Tereno S, Tremblay R, Falissard B, Guedeney A; CAPEDP Study Group. A home-visiting intervention targeting determinants of infant mental health: the study protocol for the CAPEDP randomized controlled trial in France. BMC Public Health. 2012 Aug 13;12:648. doi: 10.1186/1471-2458-12-648. PMID 22888979